CLINICAL TRIAL: NCT04500977
Title: Womens Leadership Intervention Program
Brief Title: Training Health Promotion Women Community Leaders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Jerusalem Municipality (Unknown)
Responsible Party: Principal Investigator, Donna R Zwas, Director of Linda Joy Pollin Cardiovascular Wellness Center for Women, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LDSP-HMO-CTIL
Record Dates: First submitted 2020-03-01; First posted 2020-08-06 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Sedentary Behavior; Risk Reduction
MeSH Terms: conditions — Sedentary Behavior; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Training of community members in leadership and community-based health promotion skills
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training community health promotion leaderss (Experimental): Community women are trained in leadership and community-based health promotion skills
  Interventions: Behavioral: leadership empowerment

INTERVENTIONS:
Behavioral: leadership empowerment — In the leadership program, women were taught more about the manner in which to bring about a change in one's health by adapting a healthy life style, leadership and facilitation skills and the development, implementation and evaluation process required to conduct a community program that will impact society. Women learned how to map needs and resources, define goals and objectives, develop, implement and evaluate a community based program.

SUMMARY:
Goal of the Program:

To develop personal and group ability for participants in the DPP to plan and implement health promotion programs.

Objectives:

1. Develop skills in the planning, implementation, and assessment of community-based health promotion programs
2. Personal, group and community capacity development in health promotion

DETAILED DESCRIPTION:
All participants were graduates of our previously implemented diabetes prevention program (DPP), in which women learned the health dangers involved in a sendentary life style, and unhealthy diet, a lack of planned physical activity, insufficient personal health management, and smoking. The importacne of adopting a healthy lifestyle, and how to achieve this goal was stressed. The 24 graduates most motivated to empower others were chosen to take part in this 12 session leadership program. In the leadership program, women were taught more about the manner in which to bring about a change in one's health by adopting a healthy lifestyle, leadership, and facilitation skills and the development, implementation, and evaluation process required to conduct a community program that will impact society as a whole. Women learned how to map needs and resources, define goals and objectives, implement and evaluate a community based program. Following frontal training, three action grousp were established. Each group was responsible for developing and implementing a program in the community. Programs based on initiatives set during the first stage of the DPP included: working in schools to promote a healthy lifestyle, community work targeting non-working/homemaker women ages 25+, enhancing physical activity in the community, and empowering teens. Together, all of these initiatives: increased awareness of fast food dangers, increased awareness to the dangers of nargillah smoking, and increased awareness as to the importance of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* had to previously take part in the previously implemented diabetes prevention program (DPP)
* had to have interest and ability in developing programs

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — As per self-identification
Enrollment: 150 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Program implementation | 12 months after completion of the course
  Three programs will be implemented by the group within 12 months of initiation of the course.
RE-AIM assessment of intervention quality | 12 months after completion of the course
  The RE-AIM assessment tool assesses Reach, Effectiveness, Adoption, Implementation, and Maintenance of the intervention programs. Each domain is assessed by questions adapted from the RE-AIM framework. Each item is scored as fully implemented, partially implemented or not implemented, with 0 as not, 0.5 as partially and 1.0 as fully, The questions for each item are averaged for a score that ranges from 0-1, with one being full implementation

SECONDARY OUTCOMES:
health promotion leadership self efficacy | upon completion of the course, approximately 14 weeks after initiating the intervention.
  13 item questionnaire with scores ranging from 13- 52, with 52 representing higher self efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Donna Zwas, MD MPH, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No
deidentified data may be shared upon reasonable investigator request